CLINICAL TRIAL: NCT02175758
Title: A Phase 2, Open-Label, Multicenter, Multi-cohort, Single-Arm Study to Investigate the Safety and Efficacy of Sofosbuvir + Ribavirin in Adolescents and Children With Genotype 2 or 3 Chronic HCV Infection
Brief Title: Safety and Efficacy of Sofosbuvir + Ribavirin in Adolescents and Children With Genotype 2 or 3 Chronic HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-1112; 2014-002283-32 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 12 to < 18 Years Old, SOF+RBV 12 Weeks (GT 2) (Experimental): Participants between 12 to < 18 years of age with genotype (GT) 2 HCV infection weighing ≥ 45 kg will receive SOF (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules based on swallowability assessment during screening) plus RBV (up to 1400 mg) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- 12 to < 18 Years Old, SOF+RBV 24 Weeks (GT 3) (Experimental): Participants between 12 to < 18 years of age with genotype 3 HCV infection weighing ≥ 45 kg will receive SOF (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules based on swallowability assessment during screening) plus RBV (up to 1400 mg) for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV
- 6 to < 12 Years Old, SOF+RBV 12 Weeks (GT 2) (Experimental): Participants between 6 to < 12 years of age with genotype 2 HCV infection weighing ≥ 17 kg and < 45 kg will receive SOF (2 x 100 mg tablets or 4 x 50 mg oral granules based on swallowability assessment during screening) plus RBV (up to 1400 mg) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- 6 to <12 Years Old, SOF+RBV 24 Weeks (GT 3) (Experimental): Participants between 6 to < 12 years of age with genotype 3 HCV infection weighing ≥ 17 kg and < 45 kg will receive SOF (2 x 100 mg tablets or 4 x 50 mg oral granules based on swallowability assessment during screening) plus RBV (up to 1400 mg) for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV
- 3 to < 6 Years Old, SOF+RBV 12 Weeks (GT 2) (Experimental): Participants between 3 to < 6 years of age with genotype 2 HCV infection weighing ≥ 17kg will receive SOF (4 x 50 mg oral granules) plus RBV (up to 1400 mg) for 12 weeks and those weighing < 17 kg will receive SOF (3 x 50 mg oral granules) + RBV (up to 1400 mg) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- 3 to < 6 Years Old, SOF+RBV 24 Weeks (GT 3) (Experimental): Participants between 3 to < 6 years of age with genotype 2 HCV infection weighing ≥ 17kg will receive SOF (4 x 50 mg oral granules) plus RBV (up to 1400 mg) for 24 weeks and those weighing < 17 kg will receive SOF (3 x 50 mg oral granules) + RBV (up to 1400 mg) for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — SOF administered orally once daily
  Other Names: Sovaldi®; GS-7977
Drug: RBV — RBV oral solution or capsules will be administered orally in a divided daily dose based on weight
  Other Names: REBETOL®

SUMMARY:
This study will have two parts as follows:

The PK Lead-in Phase of the study will evaluate the steady state pharmacokinetics (PK) and confirm the dose of sofosbuvir (SOF) in hepatitis C virus (HCV)-infected pediatric participants. The PK Lead-in Phase will also evaluate the safety and tolerability of 7 days of dosing of SOF+ribavirin (RBV) in HCV-infected pediatric participants.

The Treatment Phase will be initiated by age cohort after confirmation of age-appropriate SOF dosage levels. Participants from the PK Lead-in Phase will immediately rollover into the Treatment Phase with no interruption of study drug administration. The Treatment Phase will evaluate the antiviral efficacy, safety, and tolerability of SOF+RBV for 12 or 24 weeks in pediatric participants with genotype 2 or 3 HCV infection, respectively.

ELIGIBILITY:
Key Inclusion Criteria:

* Consent of parent or legal guardian required
* Chronic HCV infection genotype 2 or 3
* Screening laboratory values within defined thresholds
* PK Lead-in only: all individuals must be treatment naive

Key Exclusion Criteria:

* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Co-infection with HIV, acute hepatitis A virus, or hepatitis B virus
* Clinical hepatic decompensation (ie, ascites, encephalopathy or variceal hemorrhage)
* Pregnant or nursing females
* Known hypersensitivity to study medication
* Use of any prohibited concomitant medications as within 28 days of the Day 1 visit

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (37):
- United States (16):
  - Los Angeles, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Seattle, Washington
  - Morgantown, West Virginia
- Australia (3):
  - Westmead, New South Wales
  - Melbourne, Victoria
  - New Lambton Heights
- Brussels, Belgium
- Germany (2):
  - Wuppertal, North Rhine-Westphalia
  - Berlin
- Italy (6):
  - Bologna
  - Florence
  - Milan
  - Padua
  - San Giovanni Rotondo
  - Torino
- Auckland, New Zealand
- Russia (5):
  - Saint Petersburg, Russian Federation
  - Moscow
  - Novokuznetsk
  - Saint Petersburg
  - Tolyatti
- United Kingdom (3):
  - Birmingham
  - Leeds
  - London

REFERENCES:
- [Result] Kirby B, German P, Kanwar B, Ni L, Lakatos I, Ling J, Mathias A. Pharmacokinetics of Once-Daily Sofosbuvir and Ledipasvir/Sofosbuvir in HCV-Infected Adolescents [Poster 1707]. American Association for the Study of Liver Diseases (AASLD); 2015 November 13-17, San Francisco, USA. Hepatology 2015;62 (S1): 1040A-1041A
- [Result] Garrison KL, Mathias A, Kersey K, Kanwar B, Ni L, Jain A, et al. Pharmacokinetics of Once-Daily Sofosbuvir and Ledipasvir/Sofosbuvir in HCV-Infected Pediatrics Aged 6 to <12 Years Old [Poster 878]. American Association for the Study of Liver Diseases (AASLD); 2016 11-15 November; Boston, MA. Hepatology 2016;64 (S1): 436A
- [Result] Schwarz KB, Rosenthal P, Gonzales-Peralta RP, Jonas MM, Balistreri WF, Lin CH, et al. Sofosbuvir + Ribavirin for 12 or 24 Weeks Is Safe and Effective in Adolescents with Genotype 2 or Genotype 3 Chronic Hepatitis C Infection. Hepatology 2016; 63 (Suppl 1): abstract 706.
- [Result] Wirth S, Rosenthal P, Gonzalez-Peralta RP, Jonas MM, Balistreri WF, Lin CH, Hardikar W, Kersey K, Massetto B, Kanwar B, Brainard DM, Shao J, Svarovskaia E, Kirby B, Arnon R, Murray KF, Schwarz KB. Sofosbuvir and ribavirin in adolescents 12-17 years old with hepatitis C virus genotype 2 or 3 infection. Hepatology. 2017 Oct;66(4):1102-1110. doi: 10.1002/hep.29278. Epub 2017 Aug 26. PMID 28543053
- [Result] Younossi ZM, Stepanova M, Schwarz KB, Wirth S, Rosenthal P, Gonzalez-Peralta R, Murray K, Henry L, Hunt S. Quality of life in adolescents with hepatitis C treated with sofosbuvir and ribavirin. J Viral Hepat. 2018 Apr;25(4):354-362. doi: 10.1111/jvh.12830. Epub 2017 Dec 26. PMID 29193603
- [Result] Rosenthal P, Schwarz KB, Gonzales-Peralta RP, Lin CH, Kelly DA, Nightingale S, et al. Sofosbuvir + Ribavirin for 12 or 24 Weeks Is Safe and Effective in Children 3 to <12 Years Old with Genotype 2 or Genotype 3 Chronic Hepatitis C Infection. Hepatology 2018; 68 (Suppl 1): abstract 1844.
- [Derived] Rosenthal P, Schwarz KB, Gonzalez-Peralta RP, Lin CH, Kelly DA, Nightingale S, Balistreri WF, Bansal S, Jonas MM, Massetto B, Brainard DM, Hsueh CH, Shao J, Parhy B, Davison S, Feiterna-Sperling C, Gillis LA, Indolfi G, Sokal EM, Murray KF, Wirth S. Sofosbuvir and Ribavirin Therapy for Children Aged 3 to <12 Years With Hepatitis C Virus Genotype 2 or 3 Infection. Hepatology. 2020 Jan;71(1):31-43. doi: 10.1002/hep.30821. Epub 2019 Aug 13. PMID 31222783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Europe, Russia, New Zealand, and the United States. The first participant was screened on 07 July 2014. The last study visit occurred on 13 September 2018.
Pre-assignment Details: 135 participants were screened.
Groups:
- 12 to < 18 Years Old - SOF+RBV 12 Weeks: Participants 12 to < 18 years of age with hepatitis C virus (HCV) genotype 2 received sofosbuvir (SOF) 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + ribavirin (RBV) capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks. Participants participating in the Pharmacokinetic (PK) Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
- 12 to < 18 Years Old - SOF+RBV 24 Weeks: Participants 12 to < 18 years of age with HCV genotype 3 received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
- 6 to < 12 Years Old - SOF+RBV 12 Weeks: Participants 6 to < 12 years of age with HCV genotype 2 received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
- 6 to < 12 Years Old - SOF+RBV 24 Weeks: Participants 6 to < 12 years of age with HCV genotype 3 received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
- 3 to < 6 Years Old - SOF+RBV 12 Weeks: Participants 3 to < 6 years of age with HCV genotype 2 received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
- 3 to < 6 Years Old - SOF+RBV 24 Weeks: Participants 3 to < 6 years of age with HCV genotype 3 received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
Period: PK Lead-in Phase
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Started | 4 | 6 | 2 | 10 | 4 | 8
Completed | 4 | 6 | 2 | 10 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Started | 13 (9 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 39 (33 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 13 (11 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 28 (18 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 5 (1 participant enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 8
Completed | 13 | 38 | 13 | 28 | 4 | 8
Not Completed | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- 12 to < 18 Years Old - SOF+RBV 12 Weeks: Participants 12 to < 18 years of age with HCV genotype 2 received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks.
- 12 to < 18 Years Old - SOF+RBV 24 Weeks: Participants 12 to < 18 years of age with HCV genotype 3 received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks.
- 6 to < 12 Years Old - SOF+RBV 12 Weeks: Participants 6 to < 12 years of age with HCV genotype 2 received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks.
- 6 to < 12 Years Old - SOF+RBV 24 Weeks: Participants 6 to < 12 years of age with HCV genotype 3 received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks.
- 3 to < 6 Years Old - SOF+RBV 12 Weeks: Participants 3 to < 6 years of age with HCV genotype 2 received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks.
- 3 to < 6 Years Old - SOF+RBV 24 Weeks: Participants 3 to < 6 years of age with HCV genotype 3 received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks | Total
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.9) | 15 (1.9) | 8 (2.1) | 9 (1.7) | 4 (0.8) | 5 (0.8) | 11 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 16 | 10 | 20 | 4 | 6 | 61
  Male | 8 | 23 | 3 | 8 | 1 | 2 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4 | 1 | 0 | 9
  Not Hispanic or Latino | 13 | 36 | 11 | 23 | 4 | 8 | 95
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 11 | 36 | 9 | 20 | 3 | 6 | 85
  Race: Asian | 0 | 1 | 2 | 6 | 0 | 1 | 10
  Race: Other | 0 | 1 | 2 | 2 | 1 | 1 | 7
  Race: Black or African American | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Race: Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Belgium | 0 | 0 | 1 | 1 | 0 | 0 | 2
  United States | 8 | 11 | 8 | 10 | 4 | 5 | 46
  Italy | 3 | 4 | 2 | 1 | 0 | 1 | 11
  United Kingdom | 0 | 2 | 1 | 7 | 1 | 1 | 12
  Australia | 0 | 2 | 1 | 5 | 0 | 1 | 9
  Germany | 0 | 4 | 0 | 3 | 0 | 0 | 7
  Russia | 2 | 15 | 0 | 0 | 0 | 0 | 17
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 5 | 13 | 7 | 15 | 2 | 8 | 50
  ≥ 800,000 IU/mL | 8 | 26 | 6 | 13 | 3 | 0 | 56

OUTCOME MEASURES:

1. Primary Outcome: For Participants in the PK Lead-in Phase, Pharmacokinetic (PK) Parameter: AUCtau of GS-331007 (Metabolite of SOF)
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: 6 to < 18 years of age: predose, 0.5, 1, 2, 3, 4, 8, and 12 hours postdose on Day 7; 3 to < 6 years of age: predose, 2, 4, 8, and 12 hours postdose on Day 7
Population: Intensive PK Analysis Set included all participants in the PK lead-in phase who received at least 1 dose of study drug and for whom at least 1 nonmissing PK concentration value, during the intensive sampling period, was reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- PK Lead-in: 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks: Participants 12 to < 18 years of age received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- PK Lead-in: 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks: Participants 6 to < 12 years of age received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- PK Lead-in: 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks: Participants 3 to < 6 years of age received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
Arm/Group | PK Lead-in: 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks | PK Lead-in: 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks | PK Lead-in: 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks
Number analyzed (Participants) | 10 | 10 | 10
h*ng/mL | 9106.0 (2601.96) | 7651.2 (1723.32) | 10293.7 (1860.57)
Statistical Analysis 1: Comparison: PK Lead-in: 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks; AUCtau of GS-331007 for the 12 to < 18 Years old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — Equivalence was determined if the 90% confidence intervals (CI) were within the predefined equivalence boundaries of 50% to 200% for all age groups; Percentage Geometric Mean Ratio = 129.48, 90% CI 2-sided [109.96 to 152.48]
Statistical Analysis 2: Comparison: PK Lead-in: 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks; AUCtau of GS-331007 for the 6 to < 12 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — Equivalence was determined if the 90% CIs were within the predefined equivalence boundaries of 50% to 200% for all age groups; Percentage Geometric Mean Ratio = 109.80, 90% CI 2-sided [93.25 to 129.29]
Statistical Analysis 3: Comparison: PK Lead-in: 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks; AUCtau of GS-331007 for the 3 to < 6 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 149.67, 90% CI 2-sided [127.12 to 176.21]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event During the PK Lead-in Phase or the Treatment Phase
Time Frame: Up to 24 weeks
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
percentage of participants | 0 | 0 | 0 | 0 | 20.0 | 0

3. Primary Outcome: For the Treatment Phase, Percentage of Participants With SVR at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 12 to < 18 Years Old (Total) - SOF+RBV 12 or 24 Weeks: Participants 12 to < 18 years of age received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- 3 to < 12 Years Old (Total) - SOF+RBV 12 or 24 Weeks: Participants 6 to < 12 years of age received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
  Participants 3 to < 6 years of age received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
Arm/Group | 12 to < 18 Years Old (Total) - SOF+RBV 12 or 24 Weeks | 3 to < 12 Years Old (Total) - SOF+RBV 12 or 24 Weeks | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 52 | 54 | 13 | 39 | 13 | 28 | 5 | 8
percentage of participants | 98.1 [89.7 to 100.0] | 98.1 [90.1 to 100.0] | 100.0 [75.3 to 100.0] | 97.4 [86.5 to 99.9] | 100.0 [75.3 to 100.0] | 100.0 [87.7 to 100.0] | 80.0 [28.4 to 99.5] | 100.0 [63.1 to 100.0]
Statistical Analysis 1: Comparison: 12 to < 18 Years Old (Total) - SOF+RBV 12 or 24 Weeks; The SVR12 rate for the 12 to < 18 Years Old group was compared with the historical SVR12 rate of 80% using a 2-sided exact 1-sample binomial test at the 0.05 significance level. If superiority was demonstrated in the 12 to < 18 Years Old group, then the SVR12 rate for participants aged 3 to < 12 years would be compared with 80% at the 0.05 significance level; Test type: Superiority; p < 0.001, 2-sided exact 1-sample binomial test
Statistical Analysis 2: Comparison: 3 to < 12 Years Old (Total) - SOF+RBV 12 or 24 Weeks; The SVR12 rate for the 3 to < 12 Years Old group was compared with the historical SVR12 rate of 80% using a 2-sided exact 1-sample binomial test at the 0.05 significance level; Test type: Superiority; p < 0.001, 2-sided exact 1-sample binomial test

4. Secondary Outcome: For Participants in the PK Lead-in Phase, Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only)
Population: Participants who were enrolled in the PK lead-in phase with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Change at Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- PK Lead-in: 12 to < 18 Years Old - SOF+RBV 12 Weeks: Participants 12 to < 18 years of age with HCV genotype 2 received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks.
- PK Lead-in: 12 to < 18 Years Old - SOF+RBV 24 Weeks: Participants 12 to < 18 years of age with HCV genotype 3 received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks.
- PK Lead-in: 6 to < 12 Years Old - SOF+RBV 12 Weeks: Participants 6 to < 12 years of age with HCV genotype 2 received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks.
- PK Lead-in: 6 to < 12 Years Old - SOF+RBV 24 Weeks: Participants 6 to < 12 years of age with HCV genotype 3 received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks.
- PK Lead-in: 3 to < 6 Years Old - SOF+RBV 12 Weeks: Participants 3 to < 6 years of age with HCV genotype 2 received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 weeks.
- PK Lead-in: 3 to < 6 Years Old - SOF+RBV 24 Weeks: Participants 3 to < 6 years of age with HCV genotype 3 received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 24 weeks.
Arm/Group | PK Lead-in: 12 to < 18 Years Old - SOF+RBV 12 Weeks | PK Lead-in: 12 to < 18 Years Old - SOF+RBV 24 Weeks | PK Lead-in: 6 to < 12 Years Old - SOF+RBV 12 Weeks | PK Lead-in: 6 to < 12 Years Old - SOF+RBV 24 Weeks | PK Lead-in: 3 to < 6 Years Old - SOF+RBV 12 Weeks | PK Lead-in: 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 4 | 6 | 2 | 10 | 4 | 8
log10 IU/mL
  Change at Week 1 | -3.98 (1.056) | -4.23 (0.765) | -3.82 (0.447) | -3.78 (1.234) | -4.12 (0.632) | -3.53 (0.347)
  Change at Week 2: number analyzed (Participants) | 4 | 6 | 2 | 9 | 4 | 8
  Change at Week 2 | -4.84 (0.743) | -4.34 (0.758) | -4.92 (0.674) | -4.56 (1.553) | -4.31 (0.846) | -3.94 (0.422)
  Change at Week 4 | -4.84 (0.743) | -4.34 (0.758) | -4.92 (0.674) | -4.60 (1.686) | -4.42 (1.006) | -3.97 (0.453)
  Change at Week 8 | -4.84 (0.743) | -4.34 (0.758) | -4.92 (0.674) | -4.61 (1.700) | -4.52 (1.177) | -3.97 (0.453)
  Change at Week 12 | -4.84 (0.743) | -4.34 (0.758) | -4.92 (0.674) | -4.61 (1.700) | -4.52 (1.177) | -3.97 (0.453)
  Change at Week 16: number analyzed (Participants) | 0 | 6 | 0 | 10 | 0 | 8
  Change at Week 16 |  | -4.34 (0.758) |  | -4.61 (1.700) |  | -3.97 (0.453)
  Change at Week 20: number analyzed (Participants) | 0 | 6 | 0 | 10 | 0 | 8
  Change at Week 20 |  | -4.34 (0.758) |  | -4.61 (1.700) |  | -3.97 (0.453)
  Change at Week 24: number analyzed (Participants) | 0 | 6 | 0 | 10 | 0 | 8
  Change at Week 24 |  | -4.34 (0.758) |  | -4.61 (1.700) |  | -3.97 (0.453)

5. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event During the PK Lead-in Phase
Time Frame: Up to Day 7
Population: Participants who were enrolled in the PK lead-in phase were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | PK Lead-in: 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks | PK Lead-in: 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks | PK Lead-in: 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks
Number analyzed (Participants) | 10 | 12 | 12
percentage of participants | 0 | 0 | 0

6. Secondary Outcome: For the Treatment Phase, Percentage of Participants With Sustained Virologic Response (SVR) at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
percentage of participants | 100.0 [75.3 to 100.0] | 100.0 [91.0 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [87.7 to 100.0] | 80.0 [28.4 to 99.5] | 100.0 [63.1 to 100.0]

7. Secondary Outcome: For the Treatment Phase, Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
percentage of participants | 100.0 [75.3 to 100.0] | 97.4 [86.5 to 99.9] | 100.0 [75.3 to 100.0] | 100.0 [87.7 to 100.0] | 80.0 [28.4 to 99.5] | 100.0 [63.1 to 100.0]

8. Secondary Outcome: For the Treatment Phase, Percentage of Participants Experiencing Viral Breakthrough
Description: Viral breakthrough was defined as having confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment.
Time Frame: Up to 24 weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: For the Treatment Phase, Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as having confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: For the Treatment Phase, Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only)
Population: Participants in the Full Analysis Set with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Change at Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 13 | 38 | 13 | 28 | 4 | 8
  Change at Week 1 | -4.25 (0.986) | -4.12 (0.733) | -4.12 (0.692) | -3.88 (0.928) | -4.12 (0.632) | -3.53 (0.347)
  Change at Week 2: number analyzed (Participants) | 13 | 39 | 13 | 27 | 4 | 8
  Change at Week 2 | -4.74 (0.980) | -4.86 (0.702) | -4.55 (0.812) | -4.51 (1.102) | -4.31 (0.846) | -3.94 (0.422)
  Change at Week 4: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 4 | -4.74 (0.980) | -5.01 (0.760) | -4.68 (0.843) | -4.56 (1.171) | -4.42 (1.006) | -3.97 (0.453)
  Change at Week 8: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 8 | -4.74 (0.980) | -5.02 (0.771) | -4.68 (0.843) | -4.54 (1.191) | -4.52 (1.177) | -3.97 (0.453)
  Change at Week 12: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 12 | -4.74 (0.980) | -5.02 (0.771) | -4.68 (0.843) | -4.57 (1.178) | -4.52 (1.177) | -3.97 (0.453)
  Change at Week 16: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Change at Week 16 |  | -5.02 (0.771) |  | -4.57 (1.178) |  | -3.97 (0.453)
  Change at Week 20: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Change at Week 20 |  | -5.02 (0.771) |  | -4.57 (1.178) |  | -3.97 (0.453)
  Change at Week 24: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Change at Week 24 |  | -5.02 (0.771) |  | -4.57 (1.178) |  | -3.97 (0.453)

11. Secondary Outcome: For the Treatment Phase, Percentage of Participants With HCV RNA < LLOQ While On Treatment
Time Frame: Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only)
Population: Participants in the Full Analysis Set with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
percentage of participants
  Week 1: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Week 1 | 30.8 [9.1 to 61.4] | 30.8 [17.0 to 47.6] | 46.2 [19.2 to 74.9] | 39.3 [21.5 to 59.4] | 50.0 [6.8 to 93.2] | 37.5 [8.5 to 75.5]
  Week 2: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Week 2 | 100.0 [75.3 to 100.0] | 74.4 [57.9 to 87.0] | 76.9 [46.2 to 95.0] | 78.6 [59.0 to 91.7] | 75.0 [19.4 to 99.4] | 87.5 [47.3 to 99.7]
  Week 4: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Week 4 | 100.0 [75.3 to 100.0] | 92.3 [79.1 to 98.4] | 100.0 [75.3 to 100.0] | 96.4 [81.7 to 99.9] | 75.0 [19.4 to 99.4] | 100.0 [63.1 to 100.0]
  Week 8: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Week 8 | 100.0 [75.3 to 100.0] | 100.0 [91.0 to 100.0] | 100.0 [75.3 to 100.0] | 96.4 [81.7 to 99.9] | 100.0 [39.8 to 100.0] | 100.0 [63.1 to 100.0]
  Week 12: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Week 12 | 100.0 [75.3 to 100.0] | 100.0 [91.0 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [87.7 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [63.1 to 100.0]
  Week 16: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Week 16 |  | 100.0 [91.0 to 100.0] |  | 100.0 [87.7 to 100.0] |  | 100.0 [63.1 to 100.0]
  Week 20: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Week 20 |  | 100.0 [91.0 to 100.0] |  | 100.0 [87.7 to 100.0] |  | 100.0 [63.1 to 100.0]
  Week 24: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Week 24 |  | 100.0 [91.0 to 100.0] |  | 100.0 [87.7 to 100.0] |  | 100.0 [63.1 to 100.0]

12. Secondary Outcome: For the Treatment Phase, Percentage of Participants With Alanine Aminotransferase (ALT) Normalization
Description: ALT normalization was defined as ALT > the upper limit of normal (ULN) at baseline and ALT ≤ ULN at each visit. One participant in the 3 to < 6 Years Old 12 Weeks group had ALT > ULN at Baseline, but had no other available data.
Time Frame: Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only), and Posttreatment Week 4
Population: Participants in the Full Analysis Set with ALT > ULN at Baseline with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Weeks 16, 20, and 24 because they were only treated for 12 weeks. One participant in the 3 to < 6 Years Old 12 Weeks group had ALT > ULN at Baseline, but had no other available data.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 4 | 22 | 4 | 16 | 0 | 2
percentage of participants
  Week 1 | 50.0 | 63.6 | 25.0 | 75.0 |  | 100.0
  Week 2: number analyzed (Participants) | 4 | 22 | 3 | 15 | 0 | 2
  Week 2 | 100.0 | 90.9 | 100.0 | 93.3 |  | 100.0
  Week 4: number analyzed (Participants) | 3 | 22 | 4 | 15 | 0 | 2
  Week 4 | 100.0 | 95.5 | 100.0 | 100.0 |  | 100.0
  Week 8: number analyzed (Participants) | 4 | 22 | 3 | 15 | 0 | 2
  Week 8 | 100.0 | 95.5 | 100.0 | 100.0 |  | 100.0
  Week 12 | 100.0 | 100.0 | 100.0 | 100.0 |  | 100.0
  Week 16: number analyzed (Participants) | 0 | 21 | 0 | 15 | 0 | 2
  Week 16 |  | 100.0 |  | 100.0 |  | 100.0
  Week 20: number analyzed (Participants) | 0 | 22 | 0 | 16 | 0 | 2
  Week 20 |  | 100.0 |  | 100.0 |  | 100.0
  Week 24: number analyzed (Participants) | 0 | 21 | 0 | 15 | 0 | 2
  Week 24 |  | 100.0 |  | 100.0 |  | 100.0
  Posttreatment Week 4: number analyzed (Participants) | 4 | 16 | 3 | 12 | 0 | 2
  Posttreatment Week 4 | 100.0 | 100.0 | 100.0 | 100.0 |  | 100.0

13. Secondary Outcome: For the Treatment Phase, Change From Baseline in Height
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only), and Posttreatment Weeks 4, 12, and 24
Population: Participants in the Safety Analysis Set with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Change at Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
centimeters
  Change at Week 1: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 1 | 0.1 (1.10) | 0.0 (0.57) | 0.0 (0.57) | 0.0 (0.73) | 0.3 (1.12) | 0.3 (0.75)
  Change at Week 2: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 2 | 0.1 (1.07) | -0.1 (0.59) | 0.1 (0.66) | 0.0 (0.54) | 0.7 (1.09) | 0.3 (0.50)
  Change at Week 4: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 4 | 0.2 (1.20) | 0.2 (0.78) | 0.3 (0.67) | 0.4 (0.74) | 0.9 (0.87) | 0.5 (0.67)
  Change at Week 8: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 8 | 0.3 (1.27) | 0.2 (0.85) | 1.0 (1.00) | 0.4 (0.62) | 0.9 (0.72) | 0.8 (0.51)
  Change at Week 12: number analyzed (Participants) | 12 | 39 | 13 | 28 | 4 | 8
  Change at Week 12 | 0.5 (1.68) | 0.3 (0.95) | 0.8 (0.81) | 0.7 (0.68) | 1.5 (0.45) | 1.7 (1.84)
  Change at Week 16: number analyzed (Participants) | 0 | 38 | 0 | 28 | 0 | 8
  Change at Week 16 |  | 0.4 (0.91) |  | 1.1 (0.93) |  | 1.8 (0.79)
  Change at Week 20: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Change at Week 20 |  | 0.5 (1.10) |  | 1.6 (1.15) |  | 2.5 (1.01)
  Change at Week 24: number analyzed (Participants) | 0 | 36 | 0 | 27 | 0 | 8
  Change at Week 24 |  | 0.8 (1.54) |  | 2.1 (0.88) |  | 2.7 (1.05)
  Change at Posttreatment Week 4: number analyzed (Participants) | 13 | 38 | 13 | 28 | 4 | 8
  Change at Posttreatment Week 4 | 0.5 (1.79) | 0.9 (1.70) | 1.4 (0.80) | 2.6 (1.17) | 1.6 (0.91) | 3.5 (0.85)
  Change at Posttreatment Week 12: number analyzed (Participants) | 12 | 38 | 13 | 28 | 4 | 8
  Change at Posttreatment Week 12 | 1.4 (1.65) | 1.3 (1.90) | 2.4 (1.02) | 3.8 (1.30) | 2.8 (1.81) | 4.0 (0.95)
  Change at Posttreatment Week 24: number analyzed (Participants) | 13 | 37 | 13 | 27 | 3 | 8
  Change at Posttreatment Week 24 | 1.6 (1.89) | 1.8 (2.83) | 4.2 (1.11) | 5.1 (1.59) | 5.0 (1.61) | 5.7 (1.27)

14. Secondary Outcome: For the Treatment Phase, Change From Baseline in Weight
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
Number analyzed (Participants) | 13 | 39 | 13 | 28 | 5 | 8
kilograms
  Change at Week 1: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 1 | -0.7 (1.28) | -0.4 (1.36) | 0.2 (0.82) | 0.0 (0.55) | 0.2 (0.10) | -0.2 (0.51)
  Change at Week 2: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 2 | -0.2 (0.87) | -0.3 (0.99) | 0.3 (1.08) | 0.0 (0.64) | 0.5 (0.21) | -0.1 (0.50)
  Change at Week 4: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 4 | -0.2 (1.67) | -0.1 (1.15) | 0.4 (0.90) | 0.1 (0.90) | 0.0 (0.22) | -0.1 (0.49)
  Change at Week 8: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 8 | -0.5 (2.39) | 0.0 (1.53) | 0.6 (1.57) | 0.1 (1.21) | 0.3 (0.14) | 0.0 (0.55)
  Change at Week 12: number analyzed (Participants) | 13 | 39 | 13 | 28 | 4 | 8
  Change at Week 12 | -0.4 (2.62) | -0.1 (2.01) | 0.9 (2.15) | 0.5 (1.35) | 0.3 (0.22) | 0.1 (0.85)
  Change at Week 16: number analyzed (Participants) | 0 | 38 | 0 | 28 | 0 | 8
  Change at Week 16 |  | 0.2 (2.35) |  | 0.6 (1.34) |  | 0.1 (0.76)
  Change at Week 20: number analyzed (Participants) | 0 | 39 | 0 | 28 | 0 | 8
  Change at Week 20 |  | 0.1 (2.65) |  | 0.9 (1.59) |  | 0.4 (0.86)
  Change at Week 24: number analyzed (Participants) | 0 | 36 | 0 | 27 | 0 | 8
  Change at Week 24 |  | 0.5 (3.13) |  | 1.2 (1.91) |  | 0.4 (1.03)
  Change at Posttreatment Week 4: number analyzed (Participants) | 13 | 38 | 13 | 28 | 4 | 8
  Change at Posttreatment Week 4 | -0.3 (3.19) | 0.9 (3.24) | 1.2 (2.20) | 1.3 (2.19) | 0.5 (0.27) | 0.7 (1.05)
  Change at Posttreatment Week 12: number analyzed (Participants) | 13 | 38 | 13 | 28 | 4 | 8
  Change at Posttreatment Week 12 | 0.9 (2.69) | 2.1 (3.73) | 2.1 (3.28) | 2.2 (2.21) | 1.0 (0.88) | 0.9 (1.12)
  Change at Posttreatment Week 24: number analyzed (Participants) | 13 | 37 | 13 | 27 | 3 | 8
  Change at Posttreatment Week 24 | 2.5 (4.98) | 3.0 (4.62) | 3.8 (3.67) | 3.5 (2.42) | 1.3 (1.10) | 1.7 (1.28)

15. Secondary Outcome: For the Treatment Phase, Number of Male Participants With a Change From Baseline in Tanner Stage for Pubic Hair
Description: Tanner Stages is a scale that defines physical measurements of development based on external primary and secondary sex characteristics. It was used in this study to assess pubertal development with values ranging from Stage 1 (pre-pubertal characteristics) to Stage 5 (adult or mature characteristics). Any shifts (increase or decrease) in Tanner Stage from Baseline were analyzed and presented.
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Male participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks: Male participants 12 to < 18 years of age received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks: Male participants 6 to < 12 years of age received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks: Male participants 3 to < 6 years of age received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks
Number analyzed (Participants) | 31 | 11 | 3
Participants
  End of Treatment: No Change | 23 | 10 | 3
  End of Treatment: Increase | 8 | 1 | 0
  End of Treatment: Decrease | 0 | 0 | 0
  Posttreatment Week 12: number analyzed (Participants) | 30 | 11 | 3
  Posttreatment Week 12: No Change | 20 | 9 | 3
  Posttreatment Week 12: Increase | 10 | 2 | 0
  Posttreatment Week 12: Decrease | 0 | 0 | 0
  Posttreatment Week 24: No Change | 20 | 9 | 3
  Posttreatment Week 24: Increase | 11 | 2 | 0
  Posttreatment Week 24: Decrease | 0 | 0 | 0

16. Secondary Outcome: For the Treatment Phase, Number of Male Participants With a Change From Baseline in Tanner Stage for Genitalia Development
Description: as for outcome 15
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Male participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks
Number analyzed (Participants) | 31 | 11 | 3
Participants
  End of Treatment: No Change | 24 | 11 | 3
  End of Treatment: Increase | 7 | 0 | 0
  End of Treatment: Decrease | 0 | 0 | 0
  Posttreatment Week 12: number analyzed (Participants) | 30 | 11 | 3
  Posttreatment Week 12: No Change | 21 | 10 | 3
  Posttreatment Week 12: Increase | 9 | 1 | 0
  Posttreatment Week 12: Decrease | 0 | 0 | 0
  Posttreatment Week 24: No Change | 20 | 9 | 3
  Posttreatment Week 24: Increase | 11 | 2 | 0
  Posttreatment Week 24: Decrease | 0 | 0 | 0

17. Secondary Outcome: For the Treatment Phase, Number of Female Participants With a Change From Baseline in Tanner Stage for Pubic Hair
Description: as for outcome 15
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Female participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks: Female participants 12 to < 18 years of age received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks: Female participants 6 to < 12 years of age received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks: Female participants 3 to < 6 years of age received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks
Number analyzed (Participants) | 21 | 30 | 8
Participants
  End of Treatment: No Change | 20 | 24 | 8
  End of Treatment: Increase | 1 | 6 | 0
  End of Treatment: Decrease | 0 | 0 | 0
  Posttreatment Week 12: number analyzed (Participants) | 20 | 29 | 8
  Posttreatment Week 12: No Change | 18 | 23 | 8
  Posttreatment Week 12: Increase | 2 | 6 | 0
  Posttreatment Week 12: Decrease | 0 | 0 | 0
  Posttreatment Week 24: number analyzed (Participants) | 20 | 30 | 8
  Posttreatment Week 24: No Change | 18 | 22 | 8
  Posttreatment Week 24: Increase | 2 | 8 | 0
  Posttreatment Week 24: Decrease | 0 | 0 | 0

18. Secondary Outcome: For the Treatment Phase, Number of Female Participants With a Change From Baseline in Tanner Stage for Breast Development
Description: as for outcome 15
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Female participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks
Number analyzed (Participants) | 21 | 30 | 8
Participants
  End of Treatment: No Change | 20 | 24 | 8
  End of Treatment: Increase | 1 | 5 | 0
  End of Treatment: Decrease | 0 | 1 | 0
  Posttreatment Week 12: number analyzed (Participants) | 20 | 29 | 8
  Posttreatment Week 12: No Change | 17 | 24 | 8
  Posttreatment Week 12: Increase | 3 | 5 | 0
  Posttreatment Week 12: Decrease | 0 | 0 | 0
  Posttreatment Week 24: number analyzed (Participants) | 20 | 30 | 8
  Posttreatment Week 24: No Change | 16 | 19 | 8
  Posttreatment Week 24: Increase | 4 | 11 | 0
  Posttreatment Week 24: Decrease | 0 | 0 | 0

19. Secondary Outcome: For the Treatment Phase, Palatability of SOF Granules at Day 1 as Assessed by the Percentage of Participants Able/Unable to Taste the SOF Oral Granules
Description: Participants were asked if they were able to taste the SOF oral granules.
Time Frame: Day 1
Population: Participants in the Safety Analysis Set who performed the palatability assessment were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks: Participants 12 to < 18 years of age received SOF 400 mg (1 x 400 mg tablet, 4 x 100 mg tablets, or 8 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks: Participants 6 to < 12 years of age received SOF 200 mg (2 x 100 mg tablets or 4 x 50 mg oral granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
- 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks: Participants 3 to < 6 years of age received SOF (weight ≥ 17 kg: 200 mg granules; weight < 17 kg: 150 mg granules) once daily + RBV capsules or oral solution (up to 1400 mg, dose depending on weight) for 12 or 24 weeks.
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 or 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 or 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 or 24 Weeks
Number analyzed (Participants) | 1 | 7 | 12
percentage of participants
  Able to Taste SOF Granules: Yes | 0 | 42.9 | 75.0
  Able to Taste SOF Granules: No | 100.0 | 57.1 | 25.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs): First dose date up to Week 12 or 24 (depending on group) plus 30 days (includes AEs occurring during the PK Lead-in Phase); All-Cause Mortality: Up to Posttreatment Week 24
Description: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | 12 to < 18 Years Old - SOF+RBV 12 Weeks | 12 to < 18 Years Old - SOF+RBV 24 Weeks | 6 to < 12 Years Old - SOF+RBV 12 Weeks | 6 to < 12 Years Old - SOF+RBV 24 Weeks | 3 to < 6 Years Old - SOF+RBV 12 Weeks | 3 to < 6 Years Old - SOF+RBV 24 Weeks
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/39 | 0/13 | 0/28 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/39 | 0/13 | 0/28 | 0/5 | 1/8
Other Adverse Events (participants affected / at risk) | 12/13 | 27/39 | 9/13 | 24/28 | 5/5 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12 to < 18 Years Old - SOF+RBV 12 Weeks (N=13) | 12 to < 18 Years Old - SOF+RBV 24 Weeks (N=39) | 6 to < 12 Years Old - SOF+RBV 12 Weeks (N=13) | 6 to < 12 Years Old - SOF+RBV 24 Weeks (N=28) | 3 to < 6 Years Old - SOF+RBV 12 Weeks (N=5) | 3 to < 6 Years Old - SOF+RBV 24 Weeks (N=8)
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12 to < 18 Years Old - SOF+RBV 12 Weeks (N=13) | 12 to < 18 Years Old - SOF+RBV 24 Weeks (N=39) | 6 to < 12 Years Old - SOF+RBV 12 Weeks (N=13) | 6 to < 12 Years Old - SOF+RBV 24 Weeks (N=28) | 3 to < 6 Years Old - SOF+RBV 12 Weeks (N=5) | 3 to < 6 Years Old - SOF+RBV 24 Weeks (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 2 | 3
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 11 | 0 | 4 | 0 | 1
Oral contusion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 11 | 3 | 3
Asthenia (General disorders) | 1 | 5 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 4 | 3 | 5 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 4 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0
Impetigo (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1 | 4 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Product use issue (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 9 | 4 | 8 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Product taste abnormal (Product Issues) | 0 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 7 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 4 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 3 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (8):
  • Study Protocol: Original (2013-12-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/Prot_000.pdf
  • Study Protocol: Amendment 1 (2014-02-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/Prot_001.pdf
  • Study Protocol: Amendment 2 (2014-03-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/Prot_002.pdf
  • Study Protocol: Amendment 3 (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/Prot_003.pdf
  • Study Protocol: Amendment 4 (2014-11-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/Prot_004.pdf
  • Study Protocol: Amendment 5 (2015-05-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/Prot_005.pdf
  • Study Protocol: Amendment 6 (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/Prot_006.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT02175758/SAP_007.pdf